CLINICAL TRIAL: NCT06115564
Title: Microbiological Assessment of Bile in Patients Undergone to Endoscopic Retrograde Cholangiography (ERCP): the "Microbile Registry"
Acronym: Microbile
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Unità Sanitaria Locale della Romagna (Other)
Responsible Party: Principal Investigator, Carlo Fabbri, MD, Azienda Unità Sanitaria Locale della Romagna
Other Study IDs: 4549/2022
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Jaundice, Obstructive; Jaundice; Malignant; Choledocholithiasis; Biliary Stricture; Biliary Disease
MeSH Terms: conditions — Jaundice, Obstructive; Jaundice; Choledocholithiasis; Gallbladder Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of bile containing DNA of the microbial components.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a prospective evaluation of the microbial assessment in patients undergoing to ERC with naive papilla; the population includes all the indication to biliary drainage.

ELIGIBILITY:
Main inclusion criteria for patient enrollment were: ability to provide an informed consent; age >/=18 years; any benignant or malignant ERCP indication.

All subjects were excluded from the study:

* Patients who have already undergone endoscopic sphincterotomy
* Patients unable to express informed consent
* Pregnant or breastfeeding women
* Patients with anatomical post-surgical alterations of the upper gastrointestinal (GI) tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any benignant or malignant ERC indication in naive papilla
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbial assessment in patients undergoing to ERC with naive papilla | July 2022 to 2023
  Coltural assessment of the bile samples obtained pre- and post-sphincterotomy during ERC in naive papilla.

SECONDARY OUTCOMES:
MDR and sentinel germs detection | July 2022 to 2023
  Determine the presence and the prevalence of MDR organisms and sentinel germs in bile.
differences in the microbial community before and after sphincterotomy. | July 2022 to 2023
  Evaluation of differences in the microbial community before and after sphincterotomy.
Identify possible correlations between pre sphincterotomy positive biliary cultures, polymicrobial population and MDR organisms with several clinical features and with laboratory signs of acute cholangitis. | July 2022 to 2023
  Identify possible correlations between pre sphincterotomy positive biliary cultures, polymicrobial population and MDR organisms with several clinical features and with laboratory signs of acute cholangitis.
Identify potential differences in the pre sphincterotomy biliary microbial community depending on type of jaundice (benign or malignant). | July 2022 to 2023
  Identify potential differences in the pre sphincterotomy biliary microbial community depending on type of jaundice (benign or malignant).
Check the presence of a possible association between specific biliary bacterial strains and definite pancreaticobiliary disorders. | July 2022 to 2023
  Check the presence of a possible association between specific biliary bacterial strains and definite pancreaticobiliary disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Fabbri, MD, Principal Investigator — AUSL Romagna
Locations (1):
- Ospedale Morgagni-Pierantoni, Forlì, Forlì-Cesena, Italy

REFERENCES:
- [Background] Nicoletti A, Ponziani FR, Nardella E, Ianiro G, Gasbarrini A, Zileri Dal Verme L. Biliary tract microbiota: a new kid on the block of liver diseases? Eur Rev Med Pharmacol Sci. 2020 Mar;24(5):2750-2775. doi: 10.26355/eurrev_202003_20548. PMID 32196626
- [Background] Molinero N, Ruiz L, Milani C, Gutierrez-Diaz I, Sanchez B, Mangifesta M, Segura J, Cambero I, Campelo AB, Garcia-Bernardo CM, Cabrera A, Rodriguez JI, Gonzalez S, Rodriguez JM, Ventura M, Delgado S, Margolles A. The human gallbladder microbiome is related to the physiological state and the biliary metabolic profile. Microbiome. 2019 Jul 4;7(1):100. doi: 10.1186/s40168-019-0712-8. PMID 31272480
- [Background] Miura F, Okamoto K, Takada T, Strasberg SM, Asbun HJ, Pitt HA, Gomi H, Solomkin JS, Schlossberg D, Han HS, Kim MH, Hwang TL, Chen MF, Huang WS, Kiriyama S, Itoi T, Garden OJ, Liau KH, Horiguchi A, Liu KH, Su CH, Gouma DJ, Belli G, Dervenis C, Jagannath P, Chan ACW, Lau WY, Endo I, Suzuki K, Yoon YS, de Santibanes E, Gimenez ME, Jonas E, Singh H, Honda G, Asai K, Mori Y, Wada K, Higuchi R, Watanabe M, Rikiyama T, Sata N, Kano N, Umezawa A, Mukai S, Tokumura H, Hata J, Kozaka K, Iwashita Y, Hibi T, Yokoe M, Kimura T, Kitano S, Inomata M, Hirata K, Sumiyama Y, Inui K, Yamamoto M. Tokyo Guidelines 2018: initial management of acute biliary infection and flowchart for acute cholangitis. J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):31-40. doi: 10.1002/jhbp.509. Epub 2018 Jan 8. PMID 28941329
- [Background] Reiter FP, Obermeier W, Jung J, Denk G, Mahajan UM, De Toni EN, Schirra J, Mayerle J, Schulz C. Prevalence, Resistance Rates, and Risk Factors of Pathogens in Routine Bile Cultures Obtained during Endoscopic Retrograde Cholangiography. Dig Dis. 2021;39(1):42-51. doi: 10.1159/000509289. Epub 2020 Jun 10. PMID 32521535
- [Background] Chandra S, Klair JS, Soota K, Livorsi DJ, Johlin FC. Endoscopic Retrograde Cholangio-Pancreatography-Obtained Bile Culture Can Guide Antibiotic Therapy in Acute Cholangitis. Dig Dis. 2019;37(2):155-160. doi: 10.1159/000493579. Epub 2018 Oct 3. PMID 30282078
- [Background] Ye F, Shen H, Li Z, Meng F, Li L, Yang J, Chen Y, Bo X, Zhang X, Ni M. Influence of the Biliary System on Biliary Bacteria Revealed by Bacterial Communities of the Human Biliary and Upper Digestive Tracts. PLoS One. 2016 Mar 1;11(3):e0150519. doi: 10.1371/journal.pone.0150519. eCollection 2016. PMID 26930491
- [Background] Gomi H, Takada T, Hwang TL, Akazawa K, Mori R, Endo I, Miura F, Kiriyama S, Matsunaga N, Itoi T, Yokoe M, Chen MF, Jan YY, Ker CG, Wang HP, Wada K, Yamaue H, Miyazaki M, Yamamoto M. Updated comprehensive epidemiology, microbiology, and outcomes among patients with acute cholangitis. J Hepatobiliary Pancreat Sci. 2017 Jun;24(6):310-318. doi: 10.1002/jhbp.452. Epub 2017 May 26. PMID 28371094